CLINICAL TRIAL: NCT00570739
Title: Effects of Metformin HCl in Combination With Colesevelam HCl, Compared to Metformin HCl Alone, as Initial Therapy in Drug naïve Subjects With Type 2 Diabetes Mellitus, and the Effects of Colesevelam HCl on the Lipid Profile in Subjects With Pre Diabetes
Brief Title: Effects of Metformin Hydrochloride (HCl) in Combination With Colesevelam HCl, Compared to Metformin HCl Alone, in Patients With Type 2 Diabetes Mellitus and the Effects of Colesevelam HCl on Lipids and Glucose on Pre-diabetic Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Michael Jones, Sr. Director, Medical Affairs, Daiichi Sankyo, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-411; IND 68,466
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2010-07-13 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Type 2 Diabetes Mellitus; Hypercholesterolemia; Pre-diabetes
Keywords: Colesevelam; Type 2 Diabetes Mellitus; Pre-diabetes; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia; Glucose Intolerance | interventions — Metformin; Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diabetic Participants: Metformin HCl+Placebo for Colesevelam (Placebo Comparator): Participants will receive either 850 mg or 1700 mg of metformin HCl, depending on tolerability + 6 placebo tablets matching colesevelam 625 mg. Study medication is to be administered once daily for 16 weeks.
  Interventions: Drug: Metformin HCl and Colesevelam Placebo
- Diabetic participants: Metformin HCl + Colesevelam (Experimental): Participants will receive either 850 mg or 1700 mg of metformin HCl, depending on tolerability + 6 colesevelam tablets, 625 mg. Study medication is to be administered once daily for 16 weeks.
  Interventions: Drug: Metformin HCl tablets and Colesevelam tablets
- Pre-diabetic Participants: Colesevelam Placebo (Placebo Comparator): Participants will receive 6 placebo tablets matching colesevelam 625 mg. Study medication is to be administered once daily for 16 weeks.
  Interventions: Drug: Colesevelam placebo
- Pre-diabetes Participants: Colesevelam (Experimental): Participants will receive 6 colesevelam tablets, 625 mg. Study medication is to be administered once daily for 16 weeks.
  Interventions: Drug: Colesevelam

INTERVENTIONS:
Drug: Metformin HCl and Colesevelam Placebo — One or two Metformin HCl tablets 850 mg (depending on tolerability) and 6 colesevelam 625 mg placebo tablets once daily for 16 weeks
  Arms: Diabetic Participants: Metformin HCl+Placebo for Colesevelam
Drug: Metformin HCl tablets and Colesevelam tablets — One or two Metformin HCl tablets 850 mg (depending on tolerability) and 6 colesevelam 625 mg tablets once daily for 16 weeks
  Arms: Diabetic participants: Metformin HCl + Colesevelam
Drug: Colesevelam placebo — Six colesevelam 625 mg placebo tablets will be given once a day for 16 weeks
  Arms: Pre-diabetic Participants: Colesevelam Placebo
Drug: Colesevelam — Six colesevelam 625 mg tablets will be given once a day for 16 weeks.
  Arms: Pre-diabetes Participants: Colesevelam

SUMMARY:
This is a 16-week double-blind, placebo-controlled (for colesevelam hydrochloride (HCl)) study in the type 2 diabetic subjects and pre-diabetic subjects. Diabetic participants will also be treated with open label, background,metformin HCl. Two-hundred sixty subjects with type 2 diabetes (T2DM) and 200 pre-diabetic subjects are planned to be be enrolled. Qualified subjects with T2DM will be randomized 1:1 to receive metformin HCl plus colesevelam HCl or metformin HCl plus placebo matching colesevelam HCl. Qualified pre-diabetic subjects will be randomized 1:1 to receive colesevelam HCl or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 79 years, inclusive.
* HbA1C in the range of greater than or equal to 6.5 percent to small than or equal to 10.0 percent, to be enrolled in the T2DM cohort.
* 2-hour post 75 g OGTT glucose levels in the range of:

  * greater than or equal to 200 mg/dL to be enrolled in the T2DM cohort, or
  * greater than or equal to 140 to 200 mg/dL to be enrolled in the pre-diabetes cohort.
* FPG levels in the range of:

  * greater than or equal to 126 mg/dL to be enrolled in the T2DM cohort, or
  * greater than or equal to 110 to smaller than or equal to 125 mg/dL to be enrolled in the pre-diabetes cohort.
* LDL-C levels greater than or equal to 100 mg/dL.
* Drug-naïve, defined as having never received treatment for T2DM or not having received antidiabetic drug therapy during the 3 months prior to screening visit.
* Previous diagnosis of:

  * T2DM or prediabetes, to be enrolled in the respective cohorts, or
  * CHD, CVD, and/or primary hypercholesterolemia + BMI greater than or equal to 25 mg/kg2 to be screened for T2DM or pre-diabetes.
* Understanding of the study procedures and agreement to participate in the study by giving written informed consent at screening visit.
* Women may be enrolled if all 3 of the following criteria (in addition to the above criteria)are met:

  * They are not pregnant (women of childbearing potential must have a negative serum pregnancy test [serum beta human chorionic gonadotropin )] at screening visit);
  * They are not breast-feeding; and
  * They do not plan to become pregnant during the study.
* In addition to all of the above criteria, women must also meet 1 of the following 3 criteria to be enrolled:

  * They have been post-menopausal for at least 1 year; or
  * They are of childbearing potential and will practice 1 of the following methods of birth control throughout the study: oral, injectable, or implantable hormonal contraceptives; intrauterine device; diaphragm plus spermicide; or female condom plus spermicide. Methods of contraception that are not acceptable are partner's use of condoms or partner's vasectomy.

Exclusion Criteria:

* History of type 1 diabetes and/or history of acute or chronic metabolic acidosis, including diabetic ketoacidosis.
* History of chronic (requiring daily for greater than 2 months) use of insulin therapy, except for the treatment of gestational diabetes.
* Current or prior (within the past 3 months) treatment with an oral antidiabetic drug.
* Current or prior (within the past 3 months) treatment with colesevelam HCl (WelChol), colestipol, colestimide, or cholestyramine.
* History of dysphagia, swallowing disorders, or intestinal motility disorder.
* Any serious disorder, including pulmonary, hepatic, gastrointestinal (including clinically significant malabsorption), uncontrolled endocrine/metabolic, hematologic/oncologic (within the last 5 years), neurologic, and psychiatric diseases, that would interfere with the conduct of the study or interpretation of the data.
* Acute coronary syndrome (eg, myocardial infarction or unstable angina), coronary intervention (coronary artery bypass graft or percutaneous transluminal coronary angioplasty or similar procedure), congestive heart failure (requiring pharmacological treatment), or transient ischemic attack within 3 months of screening visit.
* History of pancreatitis.
* History of acquired immune deficiency syndrome or human immunodeficiency virus.
* History of drug or alcohol abuse within the past 2 years.
* Hospitalization for any cause within 14 days prior to screening visit.
* History of an allergic or toxic response to colesevelam HCl or any of its components.
* Known hypersensitivity to metformin HCl.
* Serum TG greater than or equal to 500 mg/dL.
* Body mass index (BMI) greater than 40 kg/m2 .

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jones, Study Director — DSI
Locations (31):
- United States (17):
  - Birmingham, Alabama
  - Los Gatos, California
  - Tarzana, California
  - Ocala, Florida
  - Pocatello, Idaho
  - Gary, Indiana
  - New Orleans, Louisiana
  - Olive Branch, Mississippi
  - Dundee, New York
  - West Seneca, New York
  - Statesville, North Carolina
  - Kent, Ohio
  - Marion, Ohio
  - Portland, Oregon
  - Corpus Christi, Texas
  - Dallas, Texas
  - San Antonio, Texas
- Colombia (3):
  - Barranquilla, Atlántico
  - Bogota, Cundinamarca
  - Bucaramanga, Santander Department
- India (5):
  - Mumbai, Dadar
  - Durgāpura, Jaipur
  - Bangalore, Karnataka
  - Kochi, Kerala
  - Nashik, Maharashtra
- Mexico (6):
  - Las Palmas, Chihuahua
  - Delegacion, Cuauhtemoc
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Hermosillo, Sonora
  - Mérida, Yucatán

REFERENCES:
- [Derived] Rosenstock J, Hernandez-Triana E, Handelsman Y, Misir S, Jones MR. Clinical effects of colesevelam in Hispanic subjects with primary hyperlipidemia and prediabetes. Postgrad Med. 2012 Jul;124(4):14-20. doi: 10.3810/pgm.2012.07.2564. PMID 22913890
- [Derived] Goldberg RB, Rosenson RS, Hernandez-Triana E, Misir S, Jones MR. Initial combination therapy with metformin plus colesevelam improves lipoprotein particles in patients with early type 2 diabetes mellitus. J Clin Lipidol. 2012 Jul-Aug;6(4):318-24. doi: 10.1016/j.jacl.2012.05.005. Epub 2012 May 29. PMID 22836068
- [Derived] Handelsman Y, Goldberg RB, Garvey WT, Fonseca VA, Rosenstock J, Jones MR, Lai YL, Jin X, Misir S, Nagendran S, Abby SL. Colesevelam hydrochloride to treat hypercholesterolemia and improve glycemia in prediabetes: a randomized, prospective study. Endocr Pract. 2010 Jul-Aug;16(4):617-28. doi: 10.4158/EP10129.OR. PMID 20634176
- [Derived] Rosenstock J, Fonseca VA, Garvey WT, Goldberg RB, Handelsman Y, Abby SL, Lai YL, Jin X, Misir S, Nagendran S, Jones MR. Initial combination therapy with metformin and colesevelam for achievement of glycemic and lipid goals in early type 2 diabetes. Endocr Pract. 2010 Jul-Aug;16(4):629-40. doi: 10.4158/EP10130.OR. PMID 20634175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two cohorts of participants, type 2 diabetics (T2DM) and pre-diabetics, were recruited from 07 Jan 2008 to 15 Dec 2008. The sites were located in Colombia, India, Mexico, and the USA. The sites included private physician offices, group practices, clinics, hospitals, institutes, and university centers.
Pre-assignment Details: Due to the different metabolic nature of the two groups the "Total" column under Baseline Characteristics is populated with data for the diabetic group, except where the total could be obtained by just adding the number of participants. Please note: in the outcomes section, LOCF=Last Observation carried forward
Groups:
- Type 2 Diabetes Group: Placebo + Metformin: This group received 6 matching colesevalm placebo tablets/day + open-label metformin. The dose of metformin depended on the participant's tolerability. This treatment duration was 16 weeks.
- Type 2 Diabetes Group: Colesevelam + Metformin: This group received 6 colevevelam tablets 625 mg once daily + open-label metformin once a day. The dose of metformin depended on the participant's tolerance for the drug. This treatment duration was 16 weeks.
- Pre-diabetic Group: Placebo: This group was given 6 placebo tablets once a day. They matched the colesevelam tablets. This treatment duration was 16 weeks.
- Pre-diabetic Group: Colesevelam: This group was given 6 colesevelam tablets, 625mg, once a day. This treatment duration was 16 weeks.
Period: Overall Study
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin | Pre-diabetic Group: Placebo | Pre-diabetic Group: Colesevelam
Started | 141 | 145 | 108 | 108
Completed | 120 | 124 | 92 | 96
Not Completed | 21 | 21 | 16 | 12
Not completed — Adverse Event | 8 | 6 | 2 | 2
Not completed — Lost to Follow-up | 4 | 5 | 4 | 1
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 3 | 5
Not completed — Required restricted medication | 0 | 0 | 1 | 0
Not completed — Met discontinuation criteria | 1 | 0 | 1 | 1
Not completed — Other | 0 | 2 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Pre-diabetic Group: Placebo: This group received 6 colesevelam matching placebo tablets once per day for 16 weeks
- Pre-diabetic Group: Colesevelam: This group received 6 colesevelam tablets, 625mg, once per day for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin | Pre-diabetic Group: Placebo | Pre-diabetic Group: Colesevelam | Total
Number analyzed (Participants) | 141 | 145 | 108 | 108 | 502
Age Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.11) | 52.7 (11.46) | 55.7 (11.14) | 53.3 (12.27) | 53.3 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 76 | 81 | 68 | 310
  Male | 56 | 69 | 27 | 40 | 192
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 30 | 32 | 15 | 14 | 91
  Black/African American | 1 | 3 | 1 | 1 | 6
  White | 20 | 21 | 14 | 11 | 66
  Hispanic | 90 | 89 | 78 | 82 | 339
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 17 | 16 | 93
  Mexico | 56 | 58 | 40 | 41 | 195
  Colombia | 25 | 26 | 36 | 37 | 124
  India | 30 | 31 | 15 | 14 | 90
Previously diagnosed with neither diabetes nor pre-diabetes [Number; unit: Participant] | 14 | 15 | 26 | 22 | 77
Previously diagnosed with pre-diabetes [Number; unit: Participant] | 17 | 21 | 81 | 85 | 204
Previously diagnosed with type 2 diabetes [Number; unit: Participant] | 110 | 109 | 1 | 1 | 221
Body Mass Index [Mean (Standard Deviation); unit: kg/m squared] | 29.78 (4.44) | 30.58 (4.669) | 30.82 (4.18) | 30.93 (4.89) | 30.19 (4.57)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 145.7 (37.54) | 153.4 (39.04) | 106.8 (14.80) | 104.1 (11.33) | 149.6 (38.43)
Fasting insulin [Mean (Standard Deviation); unit: uIU/mL] | 12.82 (8.44) | 13.86 (15.75) | 11.03 (5.55) | 13.12 (8.75) | 13.34 (12.66)
Glucose 2 hours after meal [Mean (Standard Deviation); unit: mg/dL] | 220.3 (58.68) | 234.7 (71.36) | 153.7 (39.81) | 153.7 (37.90) | 227.7 (65.74)
Height [Mean (Standard Deviation); unit: cm] | 160.6 (10.64) | 162.3 (9.67) | 159.1 (9.95) | 160.8 (9.96) | 161.5 (10.18)
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent] | 7.53 (0.94) | 7.76 (1.04) | 6.07 (0.45) | 6.02 (0.46) | 7.65 (1.0)
Low Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 135.5 (26.66) | 129.1 (23.08) | 136.8 (28.48) | 132.8 (23.88) | 132.2 (25.07)
Weight [Mean (Standard Deviation); unit: kg] | 77.26 (16.17) | 80.84 (15.53) | 78.18 (13.76) | 80.63 (18.02) | 79.08 (15.92)

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change in Hemoglobin A1C (HbA1C) When Given to Drug-naïve, Diabetic Subjects From Baseline to 4, 8, 12 and 16 Weeks.
Time Frame: Baseline to 4, 8, 12, and 16 weeks
Population: The number analyzed equals the full analysis set. The full analysis set included all randomized subjects who took at least 1 dose of randomized study medication, and had a baseline and at least 1 post-baseline efficacy variable measurement. This analysis set was used for the summary and analysis of all efficacy variables. LOCF was not used.
Measure: Least Squares Mean (Standard Error); unit: Percentage of change in HbA1c
Groups:
- Type 2 Diabetes Group:Placebo+Metformin: This group received 6 matching colesevelam placebo tablets/day + open-label metformin. The dose of metformin depended on the participant's tolerability. The total treatment duration was 16 weeks.
- Type 2 Diabetes Group:Colesevelam+Metformin: This group received 6 colesevelam tablets 625 mg once daily + open-label metformin once a day. The dose of metformin depended on the participant's tolerance for the drug. The total treatment duration was 16 weeks.
Arm/Group | Type 2 Diabetes Group:Placebo+Metformin | Type 2 Diabetes Group:Colesevelam+Metformin
Number analyzed (Participants) | 128 | 129
Percentage of change in HbA1c
  Baseline to 4 weeks:Pla+Met, N=128, Col+Met N=129 | -0.38 (0.044) | -0.53 (0.044)
  Baseline to 8 weeks:Pla+Met, N=123, Col+Met N=125 | -0.67 (0.055) | -0.84 (0.055)
  Baseline to 12 weeks:Pla+Met, N=115, Col+Met N=123 | -0.86 (0.062) | -1.05 (0.059)
  Baseline to 16 weeks:Pla+Met, N=118, Col+Met N=122 | -0.92 (0.064) | -1.17 (0.063)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 4 weeks; Test type: Superiority or Other; p = 0.0123, ANCOVA — P-Value is for the LS mean difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.27 to -0.03]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0201, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.33 to -0.03]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 12 weeks; Test type: Superiority or Other; p = 0.0239, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.36 to -0.03]
Statistical Analysis 4: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 16 weeks; Test type: Superiority or Other; p = 0.0046, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.42 to -0.08]

2. Secondary Outcome: Fasting Plasma Glucose When Given to Drug-naïve, Diabetic Subjects From Baseline to 4, 8, 12, and 16 Weeks
Time Frame: Baseline to 4, 8, 12, and 16 weeks
Population: The No. analyzed equals the full analysis set (FAS). The FAS included all randomized subjects who took at least 1 dose of randomized study medication, had a baseline and at least 1 post-baseline efficacy variable measurement. The FAS was used for the summary and analysis of all efficacy variables. The 16 week analyses are both LOCF and no LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Type 2 Diabetes Group: Placebo+Metformin: This group received 6 matching colesevelam placebo tablets/day + open-label metformin. The dose of metformin depended on the participant's tolerability. The total treatment duration was 16 weeks.
Arm/Group | Type 2 Diabetes Group: Placebo+Metformin | Type 2 Diabetes Group:Colesevelam+Metformin
Number analyzed (Participants) | 130 | 131
mg/dL
  baseline to 4 weeks Pla+Met N=130, Col+Met N=131 | -19.0 (2.31) | -24.0 (2.30)
  baseline to 8 weeks:Pla+Met N=122, Col+Met N=126 | -24.3 (1.97) | -27.6 (1.94)
  baseline to 12 weeks:Pla+Met N=121, Col+Met N=125 | -27.3 (2.21) | -28.4 (2.18)
  baseline to 16 weeks:Pla+Met N=119, Col+Met N=124 | -28.0 (2.21) | -30.5 (2.16)
  baseline to 16wks LOCF:Pla+Met N=137,Col+Met N=138 | -25.9 (2.19) | -28.0 (2.18)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 4 Weeks; Test type: Superiority or Other; p = 0.1112, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-11.3 to 1.2]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.2167, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-8.6 to 2.0]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 12 weeks; Test type: Superiority or Other; p = 0.7269, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-7.0 to 4.9]
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 16 weeks; Test type: Superiority or Other; p = 0.4063, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-8.4 to 3.4]
Statistical Analysis 5: Comparison: Type 2 Diabetes Group: Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 16 weeks (LOCF); Test type: Superiority or Other; p = 0.4909, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-8.0 to 3.9]

3. Secondary Outcome: Fasting Insulin When Given to Drug-naïve, Diabetic Subjects From Baseline to 4, 8, 12, and 16 Weeks
Time Frame: Baseline to 4, 8, 12, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: uIU/mL
Arm/Group | Type 2 Diabetes Group:Placebo+Metformin | Type 2 Diabetes Group:Colesevelam+Metformin
Number analyzed (Participants) | 127 | 127
uIU/mL
  Baseline to 4 weeks:Pla+Met, N=127, Col+Met N=127 | -2.124 (0.7219) | -2.427 (0.7219)
  Baseline to 8 weeks:Pla+Met, N=124, Col+Met N=126 | -1.992 (0.5407) | -3.007 (0.5376)
  Baseline to 12 weeks:Pla+Met, N=117, Col+Met N=123 | -2.204 (0.5159) | -3.708 (0.5048)
  Baseline to 16 weeks:Pla+Met, N=119, Col+Met N=124 | -2.978 (0.7379) | -2.802 (0.7217)
  Baseline to16wks LOCF:Pla+Met,N=137,Col+Met N=138 | -2.847 (0.6655) | -2.637 (0.6644)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 4 weeks; Test type: Superiority or Other; p = 0.7606, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.303, 95% CI 2-sided [-2.259 to 1.653]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 8 weeks; Test type: Superiority or Other; p = 0.1782, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -1.015, 95% CI 2-sided [-2.477 to 0.447]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 12 weeks; Test type: Superiority or Other; p = 0.0332, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -1.504, 95% CI 2-sided [-2.887 to -0.121]
Statistical Analysis 4: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 16 weeks; Test type: Superiority or Other; p = 0.8610, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.176, 95% CI 2-sided [-1.805 to 2.158]
Statistical Analysis 5: Comparison: Type 2 Diabetes Group:Placebo+Metformin vs Type 2 Diabetes Group:Colesevelam+Metformin; Baseline to 16 weeks (LOCF); Test type: Superiority or Other; p = 0.8196, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.210, 95% CI 2-sided [-1.599 to 2.019]

4. Secondary Outcome: Fasting C-Peptide Levels When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 weeks
Population: The No. analyzed = the full analysis set (FAS). The FAS included all randomized subjects who took at least 1 dose of randomized study medication, and had a baseline and at least 1 post-baseline efficacy variable measurement. The FAS was used for the summary and analysis of all efficacy variables. Results are presented for both LOCF and no LOCF.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Groups:
- Type 2 Diabetes Group: Placebo + Metformin: This group received 6 matching colesevelam placebo tablets/day + open-label metformin. The dose of metformin depended on the participant's tolerability. The total treatment duration was 16 weeks.
- Type 2 Diabetes Group: Colesevelam + Metformin: This group received 6 colesevelam tablets 625 mg once daily + open-label metformin once a day. The dose of metformin depended on the participant's tolerance for the drug. The total treatment duration was 16 weeks.
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 120 | 124
ng/mL
  Baseline to 16 Weeks | -0.295 (0.0695) | -0.449 (0.0683)
  Baseline to 16Wks LOCF Pla+Met N=133,Col+Met N=134 | -0.284 (0.0650) | -0.426 (0.0644)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 weeks; Test type: Superiority or Other; p = 0.1078, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.153, 95% CI 2-sided [-0.340 to 0.034]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 weeks (LOCF); Test type: Superiority or Other; p = 0.1146, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.141, 95% CI 2-sided [-0.317 to 0.035]

5. Secondary Outcome: 30 Minute Post-Meal Glucose Levels When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Type 2 Diabetes Group: Placebo + Metformin: This group received 6 matching colesevelam placebo tablets/day + open-label metformin. The dose of metformin depended on the participant's tolerability. The treatment duration was 16 weeks.
- Type 2 Diabetes Group: Colesevelam + Metformin: This group received 6 colesevelam tablets 625 mg once daily + open-label metformin once a day. The dose of metformin depended on the participant's tolerance for the drug. The treatment duration was 16 weeks.
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 120 | 123
mg/dL
  Baseline to 16 weeks | -33.1 (3.46) | -33.1 (3.43)
  Baseline to 16Wks LOCF Pla+Met N=133,Col+Met N=132 | -29.4 (3.44) | -30.4 (3.45)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 weeks; Test type: Superiority or Other; p = 0.9933, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-9.3 to 9.4]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 weeks LOCF; Test type: Superiority or Other; p = 0.8203, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-10.5 to 8.3]

6. Secondary Outcome: 1 Hour Post-Meal Glucose Levels When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 118 | 120
mg/dL
  Baseline to 16 Weeks | -35.0 (3.91) | -41.9 (3.88)
  Baseline to 16 Weeks LOCF:N=131 Pla; N=129 Colesev | -31.4 (3.92) | -39.1 (3.94)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 weeks; Test type: Superiority or Other; p = 0.1950, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-17.5 to 3.6]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.1583, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-18.3 to 3.0]

7. Secondary Outcome: 2 Hour Post-Meal Glucose Levels to in Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 115 | 120
mg/dL
  Baseline to 16 Weeks | -33.0 (4.11) | -38.14 (4.02)
  Baseline to 16 Weeks LOCF: Pla N=129, Met N=127 | -29.4 (4.18) | -36.2 (4.14)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.3663, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-16.1 to 6.0]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.2524, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -6.6, 95% CI 2-sided [-17.9 to 4.7]

8. Secondary Outcome: 2 Hour Post-Meal Insulin Levels When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: uIU/mL
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 116 | 118
uIU/mL
  Baseline to 16 Weeks | -11.601 (3.2794) | -10.551 (3.2370)
  Baseline to 16 Weeks LOCF: Pla N=129, Met N=127 | -8.592 (3.4395) | -10.156 (3.4399)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.8158, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 1.051, 95% CI 2-sided [-7.828 to 9.929]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.7433, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -1.565, 95% CI 2-sided [-10.966 to 7.836]

9. Secondary Outcome: 2 Hour Post-Meal C-Peptide Levels When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 117 | 121
ng/mL
  Baseline to 16 Weeks | -0.317 (0.2424) | -0.102 (0.2373)
  Baseline to 16 Weeks LOCF: Pla N=129, Met N=130 | -0.205 (0.2406) | -0.135 (0.2374)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.5161, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.215, 95% CI 2-sided [-0.437 to 0.867]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.8319, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.070, 95% CI 2-sided [-0.581 to 0.722]

10. Secondary Outcome: The Percent Change of Low Density Lipoprotein Cholesterol (LDL-C) When Given to Drug-naïve, Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of change in LDL-C
Groups:
- Type 2 Diabetes Group: Colesevelam+Metformin: This group received 6 colesevelam tablets 625 mg once daily + open-label metformin once a day. The dose of metformin depended on the participant's tolerance for the drug. The total treatment duration was 16 weeks.
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam+Metformin
Number analyzed (Participants) | 122 | 124
percentage of change in LDL-C
  Baseline to 8 Weeks | -5.83 (1.631) | -24.01 (1.614)
  Baseline to 16 Weeks: Pla N=119, Met N=124 | -4.94 (1.852) | -22.02 (1.813)
  Baseline to 16 Weeks LOCF: Pla N=137, Met N=136 | -5.11 (1.695) | -21.44 (1.700)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam+Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -18.19, 95% CI 2-sided [-22.61 to -13.76]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam+Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -17.08, 95% CI 2-sided [-22.09 to -12.08]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam+Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -16.33, 95% CI 2-sided [-20.96 to -11.69]

11. Secondary Outcome: Percent Change of Non-High Density Lipoprotein (Non-HDL) Levels When Given to Drug-naïve, Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of change in non-HDL
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 122 | 125
percentage of change in non-HDL
  Baseline to 8 Weeks | -5.79 (1.327) | -18.19 (1.316)
  Baseline to 16 Weeks: Pla N=119, Met N=124 | -5.08 (1.460) | -14.36 (1.436)
  Baseline to 16 Weeks LOCF: Pla N=137, Met N=136 | -5.38 (1.338) | -13.70 (1.346)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -12.40, 95% CI 2-sided [-15.99 to -8.81]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -9.28, 95% CI 2-sided [-13.23 to -5.34]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Week LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -8.33, 95% CI 2-sided [-11.98 to -4.67]

12. Secondary Outcome: Percent Change of High Density Lipoprotein Cholesterol(HDL-C) When Given to Drug-naïve, Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 122 | 125
Percentage of change
  Baseline to 8 Weeks | 2.98 (1.506) | 5.61 (1.488)
  Baseline to 16 Weeks: Pla N=119, Met N=124 | 7.46 (1.277) | 8.78 (1.250)
  Baseline to 16 Weeks LOCF: Pla N=137, Met N=136 | 6.58 (1.160) | 8.39 (1.165)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.2026, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Median Difference (Final Values) = 2.63, 95% CI 2-sided [-1.43 to 6.70]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.4506, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 1.32, 95% CI 2-sided [-2.12 to 4.75]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.2609, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [-1.35 to 4.97]

13. Secondary Outcome: Percent Change of Total Cholesterol (TC) When Given to Drug-naïve, Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change of TC
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 122 | 125
Percentage of change of TC
  Baseline to 8 Weeks | -4.46 (1.009) | -13.26 (1.000)
  Baseline to 16 Weeks: Pla N=119, Met=124 | -2.85 (1.217) | -9.79 (1.197)
  Baseline to 16 Weeks LOCF: Pla N=137, Met=136 | -3.22 (1.115) | -9.31 (1.121)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -8.81, 95% CI 2-sided [-11.53 to -6.08]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -6.94, 95% CI 2-sided [-10.23 to -3.66]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -6.09, 95% CI 2-sided [-9.14 to -3.05]

14. Secondary Outcome: Percent Change of Triglycerides (TG)When Given to Drug-naïve, Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percentage of change of TG
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 122 | 125
Percentage of change of TG
  Baseline to 8 Weeks | -7.39 [-11.41 to 0.58] | 1.28 [-4.48 to 5.58]
  Baseline to 16 Weeks: Pla N=119, Met N=124 | -7.12 [-25.58 to 7.32] | 8.63 [-8.74 to 36.85]
  Baseline to 16 Weeks LOCF: Pla N=137, Met N=136 | -9.55 [-24.13 to 14.40] | 8.80 [6.25 to 15.88]
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 weeks; Test type: Superiority or Other; p = 0.0171, ANCOVA — The P-Value was from the non-parametric ANCOVA stratified by country; The median difference was calculated using Hodges-Lehmann point estimate and corresponding 95% CI was constructed using the method of Moses; Mean Difference (Final Values) = 7.05, 95% CI 2-sided [-0.33 to 13.99]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — The P-Value was from the non-parametric ANCOVA stratified by country; [statistical method as in outcome 14, analysis 1]; Mean Difference (Final Values) = 17.71, 95% CI 2-sided [9.66 to 25.54]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA — The P-Value was from the non-parametric ANCOVA stratified by country; [statistical method as in outcome 14, analysis 1]; Mean Difference (Final Values) = 18.62, 95% CI 2-sided [11.18 to 25.74]

15. Secondary Outcome: Percent Change of Apolipoprotein A-1 (Apo A-1) When Given to Drug-naïve, Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change in Apo A-1
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 118 | 124
Percentage of change in Apo A-1
  Baseline to 8 Weeks | 3.30 (1.047) | 6.12 (1.027)
  Baseline to 16 Weeks: Pla N=113, Met N=120 | 4.86 (1.052) | 8.51 (1.024)
  Baseline to 16 Weeks LOCF: Pla N=133, Met N=134 | 4.02 (0.957) | 8.45 (0.953)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 weeks; Test type: Superiority or Other; p = 0.0496, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.81, 95% CI 2-sided [0.0 to 5.62]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0117, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 3.65, 95% CI 2-sided [0.82 to 6.47]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0009, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 4.43, 95% CI 2-sided [1.83 to 7.03]

16. Secondary Outcome: Percent Change of Apolipoprotein B (Apo B)When Given to Drug-naïve, Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change in Apo B
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 118 | 124
Percentage of change in Apo B
  Baseline to 8 Weeks | -4.59 (1.184) | 16.15 (1.158)
  Baseline to 16 Weeks: Pla N=113, Met N=120 | -3.89 (1.340) | -13.42 (1.307)
  Baseline to 16 Weeks LOCF: Pla N=133, Met N=134 | -4.20 (1.242) | -12.17 (1.239)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -11.56, 95% CI 2-sided [-14.74 to -8.38]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -9.53, 95% CI 2-sided [-13.14 to -5.92]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -7.97, 95% CI 2-sided [-11.35 to -4.59]

17. Secondary Outcome: Percent Change of Apolipoprotein C3 (Apo C3)When Given to Drug-naïve, Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change in Apo C3
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 122 | 125
Percentage of change in Apo C3
  Baseline to 8 Weeks | 0.01 (2.527) | 12.58 (2.495)
  Baseline to 16 Weeks: Pla N=117, Met N=120 | 4.06 (2.932) | 18.58 (2.871)
  Baseline to 16 Weeks LOCF: Pla N=136, N=136 | 2.82 (2.621) | 17.89 (2.620)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0003, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 12.57, 95% CI 2-sided [5.76 to 19.38]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0003, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 14.52, 95% CI 2-sided [6.64 to 22.40]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 15.08, 95% CI 2-sided [7.95 to 22.20]

18. Secondary Outcome: Change in the Levels of Various Lipoprotein Particles When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Groups:
- Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks; Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF): This group received 6 matching colesevelam placebo tablets/day + open-label metformin. The dose of metformin depended on the participant's tolerability. The total treatment duration was 16 weeks.
- Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF): This group received 6 colesevelam tablets 625 mg once daily + open-label metformin once a day. The dose of metformin depended on the participant's tolerance for the drug. The total treatment duration was 16 weeks.
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks | Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks | Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) | Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF)
Number analyzed (Participants) | 119 | 119 | 133 | 129
nmol/L
  Total Very Low Density Lipoprotein (VLDL) Particle | -4.03 (2.361) | 2.81 (2.355) | -3.71 (2.167) | 2.68 (2.188)
  VLDL Chylomicron Particles | -0.58 (0.554) | 1.73 (0.552) | -0.58 (0.507) | 1.76 (0.511)
  Medium VLDL Particles | -2.31 (1.496) | 4.84 (1.492) | -2.28 (1.383) | 4.85 (1.396)
  Small VLDL Particles | -1.12 (1.536) | -4.00 (1.532) | -0.83 (1.413) | -4.06 (1.426)
  Total Low Density Lipoprotein (LDL) Particles | -104.0 (27.04) | -303.3 (27.05) | -109.5 (25.49) | -295.5 (25.77)
  Intermediate Density Lipoprotein Particles | -9.6 (4.24) | -21.3 (4.24) | -8.9 (4.03) | -19.6 (4.08)
  Large LDL Particles | 52.1 (15.74) | -25.5 (15.69) | 45.1 (14.60) | -24.2 (14.73)
  Small LDL Particles | -146.9 (31.63) | -256.7 (31.63) | -145.9 (29.52) | -252.7 (29.84)
  Medium Small LDL Particles | -32.0 (7.16) | -48.2 (7.15) | -30.8 (6.72) | -46.2 (6.78)
  Very Small LDL Particles | -115.0 (24.96) | -208.7 (24.97) | -115.3 (23.31) | -206.6 (23.57)
  Total High Density Lipoprotein (HDL) Particles | 1.47 (0.352) | 2.41 (0.351) | 1.34 (0.332) | 2.35 (0.335)
  Large HDL Particles | 0.64 (0.160) | 1.09 (0.161) | 0.55 (0.153) | 1.00 (0.155)
  Medium HDL Particles | -0.19 (0.275) | 0.50 (0.274) | -0.26 (0.259) | 0.59 (0.261)
  Small HDL Particles | 1.04 (0.385) | 0.74 (0.384) | 1.05 (0.362) | 0.70 (0.366)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Total Very Low Density Lipoprotein (VLDL) Particles; Test type: Superiority or Other; p = 0.0363, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 6.84, 95% CI 2-sided [0.44 to 13.24]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Total Very Low Density Lipoprotein (VLDL) Particles; Test type: Superiority or Other; p = 0.0347, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 6.39, 95% CI 2-sided [0.46 to 12.31]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; VLDL Chylomicron Particles; Test type: Superiority or Other; p = 0.0028, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.31, 95% CI 2-sided [0.80 to 3.81]
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); VLDL Chylomicron Particles; Test type: Superiority or Other; p = 0.0010, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.34, 95% CI 2-sided [0.96 to 3.73]
Statistical Analysis 5: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Medium VLDL Particles; Test type: Superiority or Other; p = 0.0006, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 7.13, 95% CI 2-sided [3.10 to 11.21]
Statistical Analysis 6: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Medium VLDL Particles; Test type: Superiority or Other; p = 0.0003, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 7.13, 95% CI 2-sided [3.35 to 10.91]
Statistical Analysis 7: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Small VLDL Particles; Test type: Superiority or Other; p = 0.1750, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -2.88, 95% CI 2-sided [-7.04 to 1.29]
Statistical Analysis 8: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Small VLDL Particles; Test type: Superiority or Other; p = 0.1007, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -3.23, 95% CI 2-sided [-7.10 to 0.63]
Statistical Analysis 9: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Total Low Density Lipoprotein (LDL) Particles; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -199.3, 95% CI 2-sided [-272.9 to -125.8]
Statistical Analysis 10: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Total Low Density Lipoprotein (LDL) Particles; Test type: Superiority or Other; p = 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -186.1, 95% CI 2-sided [-255.9 to -116.3]
Statistical Analysis 11: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Intermediate Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.0466, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -11.7, 95% CI 2-sided [-23.3 to -0.2]
Statistical Analysis 12: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Intermediate Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.0570, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -10.7, 95% CI 2-sided [-21.8 to 0.3]
Statistical Analysis 13: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Large LDL Particles; Test type: Superiority or Other; p = 0.0004, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Net) = -77.7, 95% CI 2-sided [-120.3 to -35.0]
Statistical Analysis 14: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Large LDL Particles; Test type: Superiority or Other; p = 0.0007, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -69.3, 95% CI 2-sided [-109.2 to -29.3]
Statistical Analysis 15: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Small LDL Particles; Test type: Superiority or Other; p = 0.0124, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -109.9, 95% CI 2-sided [-195.8 to -23.9]
Statistical Analysis 16: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Small LDL Particles; Test type: Superiority or Other; p = 0.0098, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -106.8, 95% CI 2-sided [-187.6 to -26.0]
Statistical Analysis 17: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Medium Small LDL Particles; Test type: Superiority or Other; p = 0.1020, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -16.2, 95% CI 2-sided [-35.6 to 3.2]
Statistical Analysis 18: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Medium Small LDL Particles; Test type: Superiority or Other; p = 0.0997, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -15.4, 95% CI 2-sided [-33.8 to 3.0]
Statistical Analysis 19: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Very Small LDL Particles; Test type: Superiority or Other; p = 0.0069, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -93.7, 95% CI 2-sided [-161.6 to -25.9]
Statistical Analysis 20: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Very Small LDL Particles; Test type: Superiority or Other; p = 0.0052, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -91.4, 95% CI 2-sided [-155.2 to -27.5]
Statistical Analysis 21: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Total High Density Lipoprotein (HDL) Particles; Test type: Superiority or Other; p = 0.0524, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-0.01 to 1.90]
Statistical Analysis 22: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Total High Density Lipoprotein (HDL) Particles; Test type: Superiority or Other; p = 0.0301, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [0.10 to 1.91]
Statistical Analysis 23: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Large HDL Particles; Test type: Superiority or Other; p = 0.0416, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.02 to 0.89]
Statistical Analysis 24: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Large HDL Particles; Test type: Superiority or Other; p = 0.0333, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [0.04 to 0.88]
Statistical Analysis 25: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Medium HDL Particles; Test type: Superiority or Other; p = 0.0693, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-0.05 to 1.44]
Statistical Analysis 26: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Medium HDL Particles; Test type: Superiority or Other; p = 0.0187, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [0.14 to 1.56]
Statistical Analysis 27: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Small HDL Particles; Test type: Superiority or Other; p = 0.5765, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-1.34 to 0.75]
Statistical Analysis 28: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Small HDL Particles; Test type: Superiority or Other; p = 0.4762, ANCOVA — P-Value is for the LS Mean Difference between treatment group; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.35 to 0.63]

19. Secondary Outcome: Change in the Size of Various Lipoprotein Particles When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nm
Groups:
- Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks; Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF): This group received 6 matching colesevelam placebo tablets/day + open-label metformin. The dose of metformin depended on the participant's tolerability. The treatment duration was 16 weeks.
- Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF): This group received 6 colesevelam tablets 625 mg once daily + open-label metformin once a day. The dose of metformin depended on the participant's tolerance for the drug. The treatment duration was 16 weeks.
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks | Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks | Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) | Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF)
Number analyzed (Participants) | 119 | 119 | 133 | 129
nm
  Very Low Density Lipoprotein Particles | -0.80 (0.868) | 1.41 (0.866) | -1.02 (0.796) | 1.73 (0.804)
  Low Density Lipoprotein Particles | 0.20 (0.053) | 0.15 (0.053) | 0.19 (0.049) | 0.15 (0.050)
  High Density Lipoprotein Particles | 0.08 (0.023) | 0.17 (0.023) | 0.08 (0.021) | 0.17 (0.022)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Very Low Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.0652, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [-0.14 to 4.57]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Very Low Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.0137, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.74, 95% CI 2-sided [0.57 to 4.92]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; Low Density Lipoprotien Particles; Test type: Superiority or Other; p = 0.4726, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.20 to 0.09]
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); Low Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.5715, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.17 to 0.10]
Statistical Analysis 5: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks vs Type 2 Diabetes Group: Colesevelam + Metformin for 16 Weeks; High Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.0083, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [0.02 to 0.15]
Statistical Analysis 6: Comparison: Type 2 Diabetes Group: Placebo + Metformin for 16 Weeks (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin for 16 Weeks(LOCF); High Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.0022, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.03 to 0.15]

20. Secondary Outcome: Change in the Calculated Total Triglycerides When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 119 | 119
mg/dL
  Baseline to 16 Weeks | -8.5 (6.44) | 17.6 (6.43)
  Baseline to 16 Weeks LOCF: Pla N=133, Met N=129 | -9.0 (5.88) | 18.2 (5.93)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0036, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 26.0, 95% CI 2-sided [8.6 to 43.5]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0010, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 27.2, 95% CI 2-sided [11.2 to 43.3]

21. Secondary Outcome: Change in the Calculated Very Low Density Lipoprotein Triglycerides When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Description: These calculated values are reported as part of an NMR analysis. The calculations are done by LipoScience, Inc., and are proprietary.
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 119 | 119
mg/dL
  Baseline to 16 Weeks | -7.4 (6.36) | 22.4 (6.34)
  Baseline to 16 Weeks LOCF: Pla N=133, Met N= 129 | -7.9 (5.81) | 22.9 (5.86)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0008, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 29.8, 95% CI 2-sided [12.5 to 47.0]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 30.7, 95% CI 2-sided [14.9 to 46.6]

22. Secondary Outcome: Change in the Calculated High Density Lipoprotein Cholesterol When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Description: as for outcome 21
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 119 | 119
mg/dL
  Baseline to 16 Weeks | 3.2 (0.62) | 5.8 (0.62)
  Baseline to 16 Weeks LOCF: Pla N=133, Met N=129 | 2.9 (0.59) | 5.6 (0.60)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0033, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [0.9 to 4.3]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0008, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [1.2 to 4.4]

23. Primary Outcome: Percent Change of Hemoglobin A1C (HbA1C) From Baseline to 16 Weeks When Given as Initial Therapy to Drug-naïve, Diabetic Subjects.
Time Frame: Baseline to 16 weeks
Population: The number analyzed equals the full analysis set. The full analysis set included all randomized subjects who took at least 1 dose of randomized study medication, and had a baseline and at least 1 post-baseline efficacy variable measurement. This analysis set was used for the summary and analysis of all efficacy variables. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: Percentage of change of hemoglobin A1C
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 137 | 138
Percentage of change of hemoglobin A1C | -0.83 (0.064) | -1.09 (0.064)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Test type: Superiority or Other; p = 0.0035, ANCOVA — P-Value is for the LS mean difference between the treatment groups; The Ancova model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.44 to -0.09]

24. Secondary Outcome: Percent of Subjects Achieving HbA1c Goal of <7.0% at Weeks 4, 8, 12, and 16 if Baseline HbA1c Was > or = to 7.0% When Given to Drug-naïve, Diabetics
Time Frame: Baseline to 4, 8, 12, and 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 90 | 93
Percent of participants
  Baseline to 4 Weeks | 31.1 | 25.8
  Baseline to 8 Weeks: Pla N=87, Met N=91 | 47.1 | 48.4
  Baseline to 12 Weeks: Pla N=79, Met N=89 | 59.5 | 64.0
  Baseline to 16 Weeks: Pla N=83, Met N=87 | 59.0 | 72.4
  Baseline to 16 Weeks LOCF: Pla N=95, Met N=99 | 55.8 | 66.7
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 4 Weeks; Test type: Superiority or Other; p = 0.5848, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 weeks; Test type: Superiority or Other; p = 0.8147, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 12 Weeks; Test type: Superiority or Other; p = 0.4957, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0467, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 5: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0589, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 6: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0049, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.38 to 6.10]
Statistical Analysis 7: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0092, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.25 to 4.76]

25. Secondary Outcome: Percent of Subject Achieving HbA1c Goal of <6.5% at Weeks 4, 8, 12, and 16 When Given to Drug-naïve, Diabetic Subjects
Time Frame: Baseline to 4, 8, 12 and 16 weeks
Population: as for outcome 2
Measure: Number; unit: Percent of particpants
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 122 | 125
Percent of particpants
  Baseline to 4 Weeks | 9.0 | 24.8
  Baseline to 8 Weeks: Pla N=118, Met N=121 | 23.7 | 36.4
  Baseline to 12 Weeks: Pla N=110, Met N=119 | 38.2 | 51.3
  Baseline to 16 Weeks: Pla N=114, Met N=118 | 44.7 | 55.9
  Baseline to 16 Weeks LOCF: Pla N=131, Met N=134 | 41.2 | 52.2
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 4 Weeks; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel; Startified by country
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0280, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 12 Weeks; Test type: Superiority or Other; p = 0.0414, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0840, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 5: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0589, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 6: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0095, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.21 to 3.96]
Statistical Analysis 7: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0088, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.20 to 3.60]

26. Secondary Outcome: Percent of Subjects Achieving Low Density Lipoprotein-Cholesterol of <100 mg/dL at Weeks 8, 16 When Given to Drug-naïve, Diabetic Subjects
Time Frame: Baseline to Weeks 8, and 16
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 117 | 115
Percent of participants
  Baseline to 8 Weeks | 16.2 | 54.8
  Baseline to 16 Weeks: Pla N=114, Met N=116 | 17.5 | 50.0
  Baseline to 16 Weeks LOCF: Pla N=131, Met N=127 | 18.3 | 48.0
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate; Odds Ratio (OR) = 5.59, 95% CI 2-sided [2.78 to 11.23]
Statistical Analysis 5: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate; Odds Ratio (OR) = 4.80, 95% CI 2-sided [2.53 to 9.10]

27. Secondary Outcome: Percent of Subjects Achieving Low Density Lipoprotein-Cholesterol Goal of <70 mg/dL at Weeks 8, 16 When Given as to Drug-naïve, Diabetics
Time Frame: Baseline to Weeks 8, and 16
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 122 | 124
Percent of participants
  Baseline to 8 Weeks | 1.6 | 13.7
  Baseline to 16 Weeks: Pla N=119, Met N=124 | 5.0 | 12.9
  Baseline to 16 Weeks LOCF: Pla N=1137, Met N=136 | 4.4 | 12.5
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0326, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0157, Cochran-Mantel-Haenszel; Stratified by country
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0870, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.88 to 7.07]
Statistical Analysis 5: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.00439, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate; Odds Ratio (OR) = 2.86, 95% CI 2-sided [1.03 to 7.94]

28. Secondary Outcome: Change in Body Weight When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: lb
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 120 | 124
lb
  Baseline to 16 Weeks | -5.11 (0.564) | -4.91 (0.552)
  Baseline to 16 Weeks LOCF: Pla N=134, Met N=134 | -4.71 (0.523) | -4.56 (0.519)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.7959, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-1.32 to 1.72]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.8371, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-1.28 to 1.57]

29. Secondary Outcome: Change in Waist-to-Hip Ratio When Given to Drug-Naive Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 120 | 124
Ratio
  Baseline to 16 Weeks | -0.0033 (0.00329) | -0.0067 (0.00323)
  Baseline to 16 Weeks LOCF: Pla N=134, Met N=134 | -0.0030 (0.00306) | -0.0065 (0.00304)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.4584, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.0033, 95% CI 2-sided [-0.0122 to 0.0055]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.4039, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.0035, 95% CI 2-sided [-0.0118 to 0.0048]

30. Primary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol (LDL-C) in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: The No. analyzed=the full analysis set (FAS). The FAS included randomized subjects who took at least 1 dose of randomized medication, had a baseline and at least 1 post-baseline efficacy variable measurement. The FAS was used for the summary and analysis of all efficacy variables. Last Observation Carried Forward was used for 16 week analyses.
Measure: Least Squares Mean (Standard Error); unit: Percentage of change in LDL-C
Groups:
- Pre-Diabetes Group: Placebo: This group received 6 matching colesevelam placebo tablets/day. The treatment duration was 16 weeks.
- Pre-Diabetes Group: Colesevelam: This group received 6 colesevelam tablets 625 mg/day. The treatment duration was 16 weeks.
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 104 | 103
Percentage of change in LDL-C | 1.70 (2.054) | -13.89 (2.088)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -15.59, 95% CI 2-sided [-21.07 to -10.11]

31. Secondary Outcome: Change in Plasma Glucose Area Under the Curve (0 to 120 Minutes) From the Baseline Glucose Tolerance Test (GTT) to the 16 Week GTT
Time Frame: Baseline vs. 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL*hr
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 114 | 116
mg/dL*hr
  Baseline to 16 Weeks | -67.10 (6.305) | -77.56 (6.266)
  Baseline to 16 Weeks LOCF: Pla N=127, Met N=124 | -60.34 (6.460) | -71.88 (6.524)
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.2289, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -10.46, 95% CI 2-sided [-27.53 to 6.62]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.1997, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -11.54, 95% CI 2-sided [-29.22 to 6.14]

32. Secondary Outcome: Percent Change of Various Calculated Lipid Parameters When Given as Initial Therapy to Drug-naïve, Diabetic From Baseline to 16 Weeks Subjects
Description: as for outcome 21
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of change
Groups:
- Type 2 Diabetes Group: Placebo + Metformin (LOCF): This group received 6 matching colesevelam placebo tablets/day + open-label metformin. The dose of metformin depended on the participant's tolerability. The treatment duration was 16 weeks.
- Type 2 Diabetes Group:Colesevelam+Metformin(LOCF): This group received 6 colesevelam tablets 625 mg once daily + open-label metformin once a day. The dose of metformin depended on the participant's tolerance for the drug. The treatment duration was 16 weeks.
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin | Type 2 Diabetes Group: Placebo + Metformin (LOCF) | Type 2 Diabetes Group:Colesevelam+Metformin(LOCF)
Number analyzed (Participants) | 119 | 119 | 133 | 129
Percentage of change
  Calculated Total Triglycerides | 1.67 | 14.48 | 0.99 | 15.11
  Calc.Very Low Density Lipoprotein Triglycerides | 7.48 | 30.28 | 6.62 | 31.34
  Calculated High Density Lipoprotein-Cholesterol | 9.51 | 17.86 | 8.70 | 17.39
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Calculated Triglycerides; Test type: Superiority or Other; p = 0.0144, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 12.81, 95% CI 2-sided [2.57 to 23.05]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin(LOCF); Calculated Triglycerides; Test type: Superiority or Other; p = 0.0037, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 14.12, 95% CI 2-sided [4.63 to 23.61]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Calculated Very Low Density Lipoprotein Triglycerides; Test type: Superiority or Other; p = 0.0060, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 22.79, 95% CI 2-sided [6.59 to 39.00]
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin(LOCF); Calculated Very Low Density Lipoprotein Triglycerides; Test type: Superiority or Other; p = 0.0013, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 24.72, 95% CI 2-sided [9.71 to 39.73]
Statistical Analysis 5: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Calculated High Density Lipoprotein-Cholesterol; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = 8.35, 95% CI 2-sided [3.71 to 13.00]
Statistical Analysis 6: Comparison: Type 2 Diabetes Group: Placebo + Metformin (LOCF) vs Type 2 Diabetes Group:Colesevelam+Metformin(LOCF); Calculated High Density Lipoprotein-Cholesterol; Test type: Superiority or Other; p = 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 8.69, 95% CI 2-sided [4.27 to 13.11]

33. Secondary Outcome: Percent of Subjects Achieving 2-Hr. Post Meal Glucose Goal of <180 mg/dL When Given to Drug-naïve, Diabetic Subjects From Baseline to Week 16
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 85 | 89
Percent of participants
  Baseline to 16 Weeks | 41.2 | 41.6
  Baseline to 16 Weeks LOCF: Pla N=95, Met N=97 | 37.9 | 41.2
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.8804, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.63 to 2.34]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.5525, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.73 to 2.60]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.5648, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.3170, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

34. Secondary Outcome: Percent of Subjects Achieving Hs-C-Reactive Protein Goal of <2.0 mg/L When Given to Drug-naïve, Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin
Number analyzed (Participants) | 78 | 82
Percent of participants
  Baseline to 16 Weeks | 21.8 | 22.0
  Baseline to 16 Weeks LOCF: Pla N=91, Met N=90 | 19.8 | 20.0
Statistical Analysis 1: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.9008, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.66 to 4.06]
Statistical Analysis 2: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.9035, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.60 to 3.37]
Statistical Analysis 3: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.2874, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 4: Comparison: Type 2 Diabetes Group: Placebo + Metformin vs Type 2 Diabetes Group: Colesevelam + Metformin; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.4344, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

35. Secondary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol in Pre-Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 Weeks
Population: The No. analyzed=the full analysis set (FAS). The FAS included randomized subjects who took at least 1 dose of randomized medication, had a baseline and at least 1 post-baseline efficacy variable measurement. The FAS was used for the summary and analysis of all efficacy variables.
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Groups:
- Pre-Diabetes Group: Placebo: This group received 6 matching colesevelam placebo tablets/day. The total treatment duration was 16 weeks.
- Pre-Diabetes Group: Colesevelam: This group received 6 colesevelam tablets 625 mg once daily. The total treatment duration was 16 weeks.
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 98 | 98
Percentage of change
  Baseline to 8 Weeks | 1.74 (1.888) | -17.88 (1.921)
  Baseline to 16 Weeks: Pla N=92, Col N=95 | 2.39 (2.191) | -15.08 (2.209)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -19.62, 95% CI 2-sided [-24.61 to -14.63]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -17.47, 95% CI 2-sided [-23.24 to -11.69]

36. Secondary Outcome: Percent Change in Non-High Density Lipoprotein-Cholesterol in Pre-Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 98 | 98
Percentage of change
  Baseline to 8 Weeks | 1.50 (1.433) | -10.98 (1.461)
  Baseline to 16 Weeks: Pla N=92, Col N=95 | 1.20 (1.850) | -9.08 (1.867)
  Baseline to 16 Weeks LOCF: Pla N=104, Col N=103 | 0.69 (1.739) | -8.37 (1.770)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -12.47, 95% CI 2-sided [-16.26 to -8.69]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -10.28, 95% CI 2-sided [-15.15 to -5.41]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -9.06, 95% CI 2-sided [-13.69 to -4.42]

37. Secondary Outcome: Percent Change in High Density Lipoprotein-Cholesterol in Pre-Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 98 | 98
Percentage of change
  Baseline to 8 Weeks | -1.12 (1.398) | 2.85 (1.433)
  Baseline to 16 Weeks: Pla N=92, Col N=95 | 4.42 (1.580) | 3.57 (1.601)
  Baseline to 16 Weeks LOCF: Pla N=104, Col N=103 | 4.06 (1.447) | 3.56 (1.481)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0357, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 3.96, 95% CI 2-sided [0.27 to 7.66]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.6878, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-5.01 to 3.31]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.7972, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-4.37 to 3.36]

38. Secondary Outcome: Percent Change in Total Cholesterol in Pre-Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 99 | 98
Percentage of change
  Baseline to 8 Weeks | 0.77 (1.169) | -8.15 (1.206)
  Baseline to 16 Weeks: Pla N=92, Col N=95 | 1.66 (1.519) | -6.59 (1.536)
  Baseline to 16 Weeks: Pla N=104, Col N=103 | 1.22 (1.422) | -6.01 (1.452)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -8.91, 95% CI 2-sided [-12.02 to -5.80]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -8.26, 95% CI 2-sided [-12.25 to -4.26]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -7.23, 95% CI 2-sided [-11.03 to -3.44]

39. Secondary Outcome: Percent Change in Apolipoprotein A-1 in Pre-Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 96 | 95
Percentage of change
  Baseline to 8 Weeks | -.032 (1.150) | 3.18 (1.190)
  Baseline to 16 Weeks: Pla N=89, Col N=94 | 3.53 (1.312) | 5.67 (1.323)
  Baseline to 16 Weeks LOCF: Pla N=102, Col N=102 | 3.68 (1.205) | 5.46 (1.232)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0257, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 3.50, 95% CI 2-sided [0.43 to 6.57]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.2238, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.13, 95% CI 2-sided [-1.32 to 5.58]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.2763, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-1.44 to 4.99]

40. Secondary Outcome: Percent Change in Apolipoprotein B in Pre-Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 96 | 95
Percentage of change
  Baseline to 8 Weeks | 1.22 (1.435) | -8.62 (1.487)
  Baseline to 16 Weeks: Pla N=89, Col N=94 | 0.67 (1.788) | -8.00 (1.807)
  Baseline to 16 Weeks LOCF: Pla N=102, Col N=102 | 0.57 (1.648) | -7.52 (1.685)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -9.83, 95% CI 2-sided [-13.68 to -5.98]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0004, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -8.67, 95% CI 2-sided [-13.40 to -3.94]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0004, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -8.09, 95% CI 2-sided [-12.50 to -3.68]

41. Secondary Outcome: Percent Change in Apolipoprotein CIII in Pre-Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 94 | 95
Percentage of change
  Baseline to 8 Weeks | 3.91 (3.301) | 17.71 (3.043)
  Baseline to 16 Weeks: Pla N=88, Col N=91 | 9.31 (5.126) | 20.89 (5.231)
  Baseline to 16 Weeks: Pla N=100, Col N=102 | 9.38 (4.627) | 19.83 (4.611)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0007, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 13.80, 95% CI 2-sided [5.87 to 21.74]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0901, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 11.58, 95% CI 2-sided [-1.83 to 24.99]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0918, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a; Mean Difference (Final Values) = 10.45, 95% CI 2-sided [-1.71 to 22.62]

42. Secondary Outcome: Percent Change in Triglycerides in Pre-Diabetic Subjects From Baseline to 8, and 16 Weeks
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 99 | 98
Percentage of change
  Baseline to 8 Weeks | 0.00 [-6.95 to 7.69] | 16.57 [4.94 to 25.83]
  Baseline to 16 Weeks: Pla N=92, Col N=95 | -4.61 [-10.46 to 5.21] | 5.91 [-0.67 to 13.27]
  Baseline to 16 Weeks: Pla N=104, Col N=103 | -4.35 [-9.85 to 5.66] | 5.91 [0.00 to 13.17]
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0005, ANCOVA — P-Value is from the non-parametric ANCOVA stratified by country; Non-parametric; Median Difference (Final Values) = 15.78, 95% CI 2-sided [6.27 to 25.83] — The median difference was calculated using Hodges-Lehmann point estimates and corresponding 95% confidence interval was constructed using the method of Moses
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0011, ANCOVA — P-Value is from the non-parametric ANCOVA stratified by country; Non-parametric; Median Difference (Final Values) = 16.07, 95% CI 2-sided [6.33 to 26.02] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0009, ANCOVA — P-Value is from the non-parametric ANCOVA stratified by country; Non-parametric; Median Difference (Final Values) = 14.33, 95% CI 2-sided [5.11 to 23.84] — [estimate comment as in outcome 42, analysis 1]

43. Secondary Outcome: Percent Change in Hs-C-Reactive Protein in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline 16 Weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 92 | 95
Percentage of change
  Baseline to 16 Weeks | -11.04 [-34.62 to 23.79] | -13.43 [-47.53 to 26.39]
  Baseline to16 LOCF: Pla N=102, Col N=101 | -10.24 [-35.78 to 21.80] | -14.12 [-46.48 to 20.93]
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.6523, ANCOVA — P-Value was from the non-parametric ANCOVA stratified by country; Non-parametric; Median Difference (Final Values) = -3.29, 95% CI 2-sided [-17.50 to 10.32] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.3934, ANCOVA — P-Value was from the non-parametric ANCOVA stratified by country; Non-parametric; Median Difference (Final Values) = -4.38, 95% CI 2-sided [-17.51 to 8.77] — [estimate comment as in outcome 42, analysis 1]

44. Secondary Outcome: Level of Various Lipoprotein Particles in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: The No. analyzed equals the full analysis set (FAS). The FAS included all randomized subjects who took at least 1 dose of randomized study medication, had a baseline and at least 1 post-baseline efficacy variable measurement. The FAS was used for the summary and analysis of all efficacy variables. These 16 week analyses are both LOCF and no LOCF.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Groups:
- Pre-Diabetes Group: Placebo (LOCF): This group received 6 matching colesevelam placebo tablets/day. The treatment duration was 16 weeks.
- Pre-Diabetes Group: Colesevelam (LOCF): This group received 6 colesevelam tablets 625 mg/day. The treatment duration was 16 weeks.
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam | Pre-Diabetes Group: Placebo (LOCF) | Pre-Diabetes Group: Colesevelam (LOCF)
Number analyzed (Participants) | 89 | 93 | 99 | 99
nmol/L
  Total Very Low Density Lipoprotein (VLDL) Particle | 1.83 (3.363) | 1.92 (3.337) | 0.72 (3.132) | 2.25 (3.149)
  Large VLDL Chylomicron Particles | -.80 (0.459) | 1.64 (0.453) | -0.86 (0.424) | 1.53 (0.426)
  Medium VLDL Particles | 1.56 (2.004) | 6.59 (1.986) | 1.15 (1.890) | 6.40 (1.895)
  Small VLDL Particles | 1.15 (1.967) | -6.34 (1.951) | 0.52 (1.837) | -5.73 (1.844)
  Total Low Density Lipoprotein (LDL) Particles | -24.7 (38.15) | -135.2 (37.83) | -25.7 (35.97) | -138.4 (36.15)
  Intermediate Density Lipoprotein (LDL) Particles | -14.9 (5.71) | -15.3 (5.69) | -14.7 (5.37) | -17.0 (5.41)
  Large LDL Particles | 91.3 (29.20) | 27.6 (28.99) | 91.3 (26.79) | 27.5 (26.93)
  Small LDL Particles | -110.9 (44.15) | -148.6 (43.79) | -102.5 (41.72) | -149.4 (41.94)
  Medium Small LDL Particles | -22.5 (9.02) | -28.2 (8.95) | -21.5 (8.48) | -28.3 (8.52)
  Very Small LDL Particles | -78.3 (35.60) | -120.3 (35.32) | -81.0 (33.68) | -121.0 (33.86)
  Total High Density Lipoprotein (HDL) Particles | 0.30 (0.456) | 0.28 (0.452) | 0.38 (0.428) | 0.28 (0.430)
  Large HDL Particles | 0.51 (0.211) | 1.09 (0.210) | 0.53 (0.197) | 1.10 (0.198)
  Medium HDL Particles | -0.23 (0.335) | -0.03 (0.334) | -0.24 (0.310) | -0.05 (0.312)
  Small HDL Particles | 0.04 (0.475) | -0.77 (0.471) | 0.10 (0.450) | -0.75 (0.453)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Total VLDL Particles; Test type: Superiority or Other; p = 0.9838, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-8.66 to 8.84]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Total VLDL Particles; Test type: Superiority or Other; p = 0.7157, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 1.53, 95% CI 2-sided [-6.73 to 9.79]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Large VLDL Chylomicron Particles; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.44, 95% CI 2-sided [1.25 to 3.63]
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Large VLDL Chylomicron Particles; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 2.39, 95% CI 2-sided [1.27 to 3.51]
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Medium VLDL Chylomicron Particles; Test type: Superiority or Other; p = 0.0577, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 5.04, 95% CI 2-sided [-0.17 to 10.24]
Statistical Analysis 6: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Medium VLDL Chylomicron Particles; Test type: Superiority or Other; p = 0.0390, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 5.24, 95% CI 2-sided [0.27 to 10.22]
Statistical Analysis 7: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Small VLDL Particles; Test type: Superiority or Other; p = 0.0044, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -7.49, 95% CI 2-sided [-12.61 to -2.37]
Statistical Analysis 8: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Small VLDL Particles; Test type: Superiority or Other; p = 0.0118, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -6.24, 95% CI 2-sided [-11.09 to -1.40]
Statistical Analysis 9: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Total Low Density Lipoprotein (LDL) Particles; Test type: Superiority or Other; p = 0.0293, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -110.6, 95% CI 2-sided [-209.9 to -11.3]
Statistical Analysis 10: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Total Low Density Lipoprotein (LDL) Particles; Test type: Superiority or Other; p = 0.0202, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -112.7, 95% CI 2-sided [-207.6 to -17.8]
Statistical Analysis 11: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Intermediate Density Lipoprotein (LDL) Particles; Test type: Superiority or Other; p = 0.9629, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-15.2 to 14.5]
Statistical Analysis 12: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Intermediate Density Lipoprotein (LDL) Particles; Test type: Superiority or Other; p = 0.7485, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-16.5 to 11.9]
Statistical Analysis 13: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Large LDL Particles; Test type: Superiority or Other; p = 0.1007, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -63.6, 95% CI 2-sided [-139.7 to 12.5]
Statistical Analysis 14: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Large LDL Particles; Test type: Superiority or Other; p = 0.0768, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -63.8, 95% CI 2-sided [-134.6 to 6.9]
Statistical Analysis 15: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Small LDL Particles; Test type: Superiority or Other; p = 0.4143, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -47.7, 95% CI 2-sided [-162.7 to 67.3]
Statistical Analysis 16: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Small LDL Particles; Test type: Superiority or Other; p = 0.4020, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -46.9, 95% CI 2-sided [-157.1 to 63.3]
Statistical Analysis 17: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Medium Small LDL Particles; Test type: Superiority or Other; p = 0.6378, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-29.1 to 17.9]
Statistical Analysis 18: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Medium Small LDL Particles; Test type: Superiority or Other; p = 0.5528, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-29.1 to 15.6]
Statistical Analysis 19: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Very Small LDL Particles; Test type: Superiority or Other; p = 0.3730, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -42.0, 95% CI 2-sided [-134.8 to 50.8]
Statistical Analysis 20: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Very Small LDL Particles; Test type: Superiority or Other; p = 0.3764, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -40.0, 95% CI 2-sided [-129.0 to 49.0]
Statistical Analysis 21: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Total High Density Lipoprotein (HDL) Particles; Test type: Superiority or Other; p = 0.9807, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-1.20 to 1.17]
Statistical Analysis 22: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Total High Density Lipoprotein (HDL) Particles; Test type: Superiority or Other; p = 0.8615, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-1.23 to 1.03]
Statistical Analysis 23: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Large HDL Particles; Test type: Superiority or Other; p = 0.0364, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [0.04 to 1.14]
Statistical Analysis 24: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Large HDL Particles; Test type: Superiority or Other; p = 0.0340, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [0.04 to 1.08]
Statistical Analysis 25: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Medium HDL Particles; Test type: Superiority or Other; p = 0.6587, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.68 to 1.07]
Statistical Analysis 26: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Medium HDL Particles; Test type: Superiority or Other; p = 0.6554, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.63 to 1.00]
Statistical Analysis 27: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Small HDL Particles; Test type: Superiority or Other; p = 0.1957, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-2.06 to 0.42]
Statistical Analysis 28: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Small HDL Particles; Test type: Superiority or Other; p = 0.1622, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-2.03 to 0.34]

45. Secondary Outcome: Particle Size of Various Lipoprotein Particles in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam | Pre-Diabetes Group: Placebo (LOCF) | Pre-Diabetes Group: Colesevelam (LOCF)
Number analyzed (Participants) | 89 | 93 | 99 | 99
nm
  Very Low Density Lipoprotein Particles | -1.85 (0.956) | 4.15 (0.948) | -1.43 (0.877) | 3.89 (0.883)
  Low Density Lipoprotein Particles | .23 (0.068) | 0.11 (0.068) | 0.23 (0.064) | 0.12 (0.065)
  High Density Lipoprotein Particles | 0.06 (0.026) | 0.15 (0.026) | 0.05 (0.024) | 0.15 (0.024)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Very Low Density Lipoprotein Particles; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 5.99, 95% CI 2-sided [3.51 to 8.48]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Very Low Density Lipoprotein Particles; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 5.31, 95% CI 2-sided [3.00 to 7.63]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Low Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.1742, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.30 to 0.05]
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Low Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.1870, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.28 to 0.06]
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; High Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.0063, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.03 to 0.16]
Statistical Analysis 6: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); High Density Lipoprotein Particles; Test type: Superiority or Other; p = 0.0020, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [0.04 to 0.16]

46. Secondary Outcome: Change of Various Calculated Lipid Parameters in Pre-Diabetic Subjects From Baseline to 16 Weeks
Description: as for outcome 21
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam | Pre-Diabetes Group: Placebo (LOCF) | Pre-Diabetes Group: Colesevelam (LOCF)
Number analyzed (Participants) | 89 | 93 | 99 | 99
mg/dL
  Changes in Calculated Total Triglycerides | -5.0 (5.97) | 19.4 (5.91) | -6.4 (5.60) | 18.0 (5.62)
  Changes: Calculated Very Low Density Triglycerides | -4.6 (5.70) | 21.7 (5.64) | -5.9 (5.34) | 20.6 (5.36)
  Changes in Calculated High Density Lipoprotein -C | 1.4 (0.75) | 2.9 (0.74) | 1.4 (0.69) | 2.9 (0.69)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Changes in Calculated Total Triglycerides; Test type: Superiority or Other; p = 0.0022, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 24.4, 95% CI 2-sided [8.9 to 39.9]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Changes in Calculated Total Triglycerides; Test type: Superiority or Other; p = 0.0013, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 24.3, 95% CI 2-sided [9.6 to 39.1]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Changes: Calculated Very Low Density Triglycerides; Test type: Superiority or Other; p = 0.0006, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 26.3, 95% CI 2-sided [11.5 to 41.0]
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Changes: Calculated Very Low Density Triglycerides; Test type: Superiority or Other; p = 0.0003, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 26.5, 95% CI 2-sided [12.5 to 40.6]
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo; Changes in Calculated High Density Lipoprotein-Cholesterol; Test type: Superiority or Other; p = 0.1257, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.4 to 3.5]
Statistical Analysis 6: Comparison: Pre-Diabetes Group: Placebo (LOCF) vs Pre-Diabetes Group: Colesevelam (LOCF); Changes in Calculated High Density Lipoprotein-Cholesterol; Test type: Superiority or Other; p = 0.1054, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.3 to 3.3]

47. Secondary Outcome: Percent Change of HbA1c in Pre-Diabetic Subjects From Baseline to 4, 8, 12, and 16 Weeks
Time Frame: Baseline to 4, 8, 12, and 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 100 | 96
Percentage of change
  Baseline to 4 weeks | -0.06 (0.026) | -0.09 (0.028)
  Baseline to 8 weeks: Pla N=98, Col N=96 | -0.06 (0.026) | -0.10 (0.026)
  Baseline to 12 weeks: Pla N=94, Col N=94 | -0.05 (0.026) | -0.11 (0.027)
  Baseline to 16 weeks: Pla N=90, Col N=95 | -0.03 (0.034) | -0.11 (0.034)
  Baseline to 16 weeks LOCF: Pla N=106, Col N=103 | -0.03 (0.030) | -0.12 (0.031)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 4 Weeks; Test type: Superiority or Other; p = 0.2971, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.11 to 0.03]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.2567, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.11 to 0.03]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 12 Weeks; Test type: Superiority or Other; p = 0.1081, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.13 to 0.01]
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0790, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.17 to 0.01]
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0206, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.18 to -0.01]

48. Secondary Outcome: Percent Change of Fasting Plasma Glucose in Pre-Diabetic Subjects From Baseline to 4, 8, 12, and 16 Weeks
Time Frame: Baseline to 4, 8, 12, and 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 101 | 97
Percentage of change
  Baseline to 4 weeks | 0.7 (0.95) | -3.5 (0.97)
  Baseline to 8 weeks: Pla N=97, Col N=97 | -1.1 (0.94) | -3.1 (0.95)
  Baseline to 12 weeks: Pla N=95, Col N=95 | 0.4 (1.11) | -2.4 (1.13)
  Baseline to 16 weeks: Pla N=91, Col N=95 | -0.5 (1.87) | -2.8 (1.86)
  Baseline to 16 weeks LOCF: Pla N=106, Col N=103 | -0.5 (1.65) | -3.1 (1.67)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 4 Weeks; Test type: Superiority or Other; p = 0.0009, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-6.8 to -1.8]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.1184, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-4.5 to 0.5]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 12 Weeks; Test type: Superiority or Other; p = 0.0615, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-5.8 to 0.1]
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.3617, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-7.2 to 2.6]
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.2372, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-7.0 to 1.7]

49. Secondary Outcome: Percent Change of Fasting Insulin in Pre-Diabetic Subjects From Baseline to 4, 8, 12, and 16 Weeks
Time Frame: Baseline to 4, 8, 12, and 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 95 | 93
Percentage of change
  Baseline to 4 Weeks | -1.269 (0.6651) | -0.348 (0.6769)
  Baseline to 8 Weeks: Pla N=94, Col N=97 | -1.208 (0.4377) | -0.513 (0.4377)
  Baseline to 12 Weeks: Pla N=93, Col N=93 | -0.848 (0.4371) | -2.066 (0.4463)
  Baseline to 16 Weeks: Pla N=90, Col N=94 | -0.063 (1.2082) | -0.497 (1.1980)
  Baseline to 16 Weeks LOCF: Pla N=105, Col N=102 | -0.019 (1.0597) | -0.512 (1.0770)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo; Baseline to 4 Weeks; Test type: Superiority or Other; p = 0.2982, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.921, 95% CI 2-sided [-0.821 to 2.663]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.2361, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.695, 95% CI 2-sided [-0.458 to 1.848]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 12 Weeks; Test type: Superiority or Other; p = 0.0413, ANCOVA; Mean Difference (Final Values) = -1.218, 95% CI 2-sided [-2.388 to -0.049]
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.7858, ANCOVA; Mean Difference (Final Values) = -0.434, 95% CI 2-sided [-3.583 to 2.715]
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.7314, ANCOVA; Mean Difference (Final Values) = -0.493, 95% CI 2-sided [-3.321 to 2.335]

50. Secondary Outcome: Change of Fasting C-peptide Levels in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 91 | 94
ng/mL
  Baseline to 16 Weeks | 0.039 (0.1124) | -0.050 (0.1132)
  Baseline to 16 Weeks LOCF: Pla N=101, Col N=100 | 0.049 (0.1041) | -0.057 (0.1059)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.5530, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.089, 95% CI 2-sided [-0.385 to 0.207]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.4554, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.105, 95% CI 2-sided [-0.383 to 0.172]

51. Secondary Outcome: Change of Glucose Levels 30 Minutes Post Oral Glucose Tolerance Test in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 88 | 94
mg/dL
  Baseline to 16 Weeks | -0.9 (3.82) | -1.8 (3.71)
  Baseline to 16 Weeks LOCF: Pla N=96, Col N=97 | -1.3 (3.60) | -2.5 (3.58)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.8583, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-10.7 to 8.9]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.7975, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-10.5 to 8.1]

52. Secondary Outcome: Change of Glucose Levels 1 Hour Post Oral Glucose Tolerance Test in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 85 | 95
mg/dL
  Baseline to 16 Weeks | -1.0 (4.51) | -8.0 (4.33)
  Baseline to 16 Weeks LOCF: Pla N=93, Col N=98 | -0.4 (4.28) | -8.6 (4.19)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.2330, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -7.0, 95% CI [-18.5 to 4.5]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.1412, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-19.2 to 2.8]

53. Secondary Outcome: Change of Glucose Levels 2 Hours Post Oral Glucose Tolerance Test in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 90 | 95
mg/dL
  Baseline to 16 Weeks | -4.9 (4.65) | -6.3 (4.65)
  Baseline to 16 Weeks LOCF: Pla N=98, Col N=98 | -4.2 (4.40) | -6.1 (4.46)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.8192, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-13.7 to 10.8]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.7513, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-13.5 to 9.7]

54. Secondary Outcome: Change of Insulin Levels 2 Hours Post Oral Glucose Tolerance Test in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: uIU/mL
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 84 | 91
uIU/mL
  Baseline to 16 Weeks | -8.563 (6.6122) | -15.472 (6.4814)
  Baseline to 16 Weeks LOCF: Pla N=92, Col N=94 | -9.784 (6.2865) | -14.954 (6.2745)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.4301, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -6.910, 95% CI 2-sided [-24.156 to 10.336]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.5369, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -5.170, 95% CI 2-sided [-21.661 to 11.321]

55. Secondary Outcome: Change of C-Peptide Levels 2 Hours Post Oral Glucose Tolerance Test in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 85 | 93
ng/mL
  Baseline to 16 Weeks | -0.447 (0.3527) | -0.598 (0.3449)
  Baseline to 16 Weeks LOCF: Pla N=93, Col N=96 | -0.581 (0.3374) | -0.551 (0.3359)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.7447, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.151, 95% CI 2-sided [-1.068 to 0.765]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.9476, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = 0.029, 95% CI 2-sided [-0.853 to 0.911]

56. Secondary Outcome: Percent of Subjects Achieving Low Density Lipoprotein-Cholesterol of <100 mg/dL at Weeks 8, 16 in Pre-Diabetic Subjects
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 94 | 89
Percent of participants
  Baseline to 8 Weeks | 6.4 | 29.2
  Baseline to 16 Weeks: Pla N=88, Col N=86 | 10.2 | 29.1
  Baseline to 16 Weeks LOCF: Pla N=100, Col N=94 | 11.0 | 28.7
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0018, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 5.23, 95% CI 2-sided [2.06 to 13.58]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 4.46, 95% CI 2-sided [1.89 to 10.54]
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

57. Secondary Outcome: Percent of Subjects Achieving Low Density Lipoprotein-Cholesterol of <70 mg/dL at Weeks 8, 16 in Pre-Diabetic Subjects
Time Frame: Baseline to 8, and 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 98 | 98
Percent of participants
  Baseline to 8 Weeks | 2.0 | 11.2
  Baseline to 16 Weeks: Pla N=92, Col N=95 | 3.3 | 7.4
  Baseline to 16 Weeks LOCF: Pla N=104, Col N=103 | 2.9 | 6.8
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.0104, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.2224, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.53 to 9.39]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.1990, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.53 to 9.33]
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.2778, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.2785, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

58. Secondary Outcome: Change in Body Weight in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: lb
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 92 | 96
lb
  Baseline to 16 Weeks | -2.56 (0.823) | -3.24 (0.832)
  Baseline to 16 Weeks LOCF: Pla N=103, Col N=101 | -2.63 (0.758) | -3.25 (0.779)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.5353, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-2.84 to 1.48]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.5475, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-2.64 to 1.40]

59. Secondary Outcome: Change in Waist-to-Hip Ratio in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Change in Ratio
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 92 | 96
Change in Ratio
  Baseline to 16 Weeks | 0.0059 (0.00477) | -0.0058 (0.00480)
  Baseline to 16 Weeks: Pla N=103, Col N=101 | 0.0051 (0.00437) | -0.0061 (0.00447)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0678, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.0116, 95% CI 2-sided [-0.0241 to 0.0009]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0585, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -0.0112, 95% CI 2-sided [-0.0228 to 0.0004]

60. Secondary Outcome: Area Under the Curve for Plasma Glucose From 0 to 120 Minutes During the Oral Glucose Tolerance Tests in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL*hr
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 84 | 93
mg/dL*hr
  Baseline to 16 Weeks | -5.26 (6.109) | -8.27 (5.878)
  Baseline to 16 Weeks: Pla N=92, Col N=96 | -4.40 (5.791) | -9.20 (5.685)
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.7051, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-18.64 to 12.64]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.5267, ANCOVA — P-Value is for the LS Mean Difference between treatment groups; The ANCOVA model includes treatment and country as fixed effects and baseline lab value as a covariate; Mean Difference (Final Values) = -4.80, 95% CI 2-sided [-19.72 to 10.13]

61. Secondary Outcome: Percent Achievement of <140 mg/dL Plasma Glucose 2 Hours Post the Oral Glucose Tolerance Test in Pre-Diabetic Subjects Whose Corresponding Baseline Value Was >or= to 140 mg/dL From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 57 | 67
Percent of participants
  Baseline to 16 Weeks | 42.1 | 37.3
  Baseline to 16 Weeks LOCF: Pla N=61, Col N=69 | 41.0 | 37.7
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.5882, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.40 to 1.83]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.7098, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.44 to 1.96]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.6835, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.8461, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

62. Secondary Outcome: Percent Achievement of <110 mg/dL Fasting Plasma Glucose in Pre-Diabetic Subjects Whose Corresponding Baseline Value Was > or = to 110 mg/dL From Baseline to 4, 8, 12, and 16 Weeks
Time Frame: Baseline to 4, 8, 12, and 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 34 | 26
Percent of participants
  Baseline to 4 Weeks | 38.2 | 57.7
  Baseline to 8 Weeks: Pla N=34, Col N=26 | 50.0 | 42.3
  Baseline to 12 Weeks: Pla N=34, Col N=26 | 55.9 | 53.8
  Baseline to 16 Weeks: Pla N=32, Col N=25 | 56.3 | 44.0
  Baseline to 16 Weeks LOCF: Pla N=36, Col N=29 | 55.6 | 48.3
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 4 Weeks; Test type: Superiority or Other; p = 0.2079, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.4053, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 12 Weeks; Test type: Superiority or Other; p = 0.5752, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.7994, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.25 to 2.29]
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.9960, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.32 to 3.03]
Statistical Analysis 6: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.7783, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 7: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.9774, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

63. Secondary Outcome: Percent Achievement of <100 mg/dL Fasting Plasma Glucose in Pre-Diabetic Subjects Whose Corresponding Baseline Value Was > or = to 100 mg/dL From Baseline to 4, 8, 12 and 16 Weeks
Time Frame: Baseline to 4, 8, 12 and 16 weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 69 | 63
Percent of participants
  Baseline to 4 Weeks | 7.2 | 39.7
  Baseline to 8 Weeks: Pla N=68, Col N=64 | 22.1 | 29.7
  Baseline to 12 Weeks: Pla N=66, Col N=65 | 16.7 | 33.8
  Baseline to 16 Weeks: Pla N=62, Col N=64 | 27.4 | 40.6
  Baseline to 16 Weeks LOCF: Pla N=73, Col N=68 | 23.3 | 39.7
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 4 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 8 Weeks; Test type: Superiority or Other; p = 0.4058, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 12 Weeks; Test type: Superiority or Other; p = 0.0254, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.1499, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.74 to 3.55]
Statistical Analysis 5: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0420, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.97 to 4.45]
Statistical Analysis 6: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.2240, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 7: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.0593, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

64. Secondary Outcome: Percent Achievement of <140 mg/dL Plasma Glucose Post 2 Hour Glucose Tolerance Test and Fasting Plasma Glucose <110 mg/dL in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 65 | 72
Percent of participants
  Baseline to 16 Weeks | 36.9 | 30.6
  Baseline to 16 Weeks LOCF: Pla N=69, Col N=75 | 36.2 | 32.0
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.4794, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.31 to 1.40]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.6667, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.37 to 1.55]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.2768, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.4395, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

65. Secondary Outcome: Percent Achievement of Hs-C-Reactive Protein <2.0 mg/L in Pre-Diabetic Subjects Whose Corresponding Baseline Value Was > or = to 2.0 mg/L From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 69 | 60
Percent of participants
  Baseline to 16 Weeks | 13.0 | 21.7
  Baseline to 16 Weeks LOCF: Pla N=78, Col N=65 | 12.8 | 20.8
Statistical Analysis 1: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.1375, Cochran-Mantel-Haenszel — P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.89 to 6.64]
Statistical Analysis 2: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.1996, Cochran-Mantel-Haenszel; P-Value for comparing percentages was from the Cochran-Mantel-Haenszel test stratified by country; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.85 to 5.82]
Statistical Analysis 3: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks; Test type: Superiority or Other; p = 0.0829, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate
Statistical Analysis 4: Comparison: Pre-Diabetes Group: Placebo vs Pre-Diabetes Group: Colesevelam; Baseline to 16 Weeks LOCF; Test type: Superiority or Other; p = 0.1037, Regression, Logistic; Contained treatment and country as factors and baseline lab value as a covariate

66. Secondary Outcome: Percent of Subjects Meeting Type 2 Diabetes Criteria (Fasting Plasma Glucose >or= to 126 mg/dL or Plasma Glucose >or= to 200 mg/dL Post 2 Hr Glucose Tolerance Test in Pre-Diabetic Subjects From Baseline to 16 Weeks
Time Frame: Baseline to 16 Weeks
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Pre-Diabetes Group: Placebo | Pre-Diabetes Group: Colesevelam
Number analyzed (Participants) | 79 | 81
Percent of participants
  Baseline to 16 Weeks | 10.1 | 11.1
  Baseline to 16 Weeks LOCF: Pla N=87, Col N=84 | 10.3 | 10.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of the informed consent form until the end of the study + a follow up period (until the AE resolved or stabilized). This period of time equals about 17.5 weeks.
Description: AEs were noted by investigator or reported by subject. Nature, duration, remedial action, and severity of AE were recorded. Lab abnormalities were AEs if they needed intervention, further investigation, led to a change in medication, or were part of a larger disease process. Only 107 in the prediabetes colesevelam group because 1 did not take drug.
Arm/Group | Type 2 Diabetes Group: Placebo + Metformin | Type 2 Diabetes Group: Colesevelam + Metformin | Pre-diabetic Group: Placebo | Pre-diabetic Group: Colesevelam
Serious Adverse Events (participants affected / at risk) | 1/141 | 2/145 | 2/108 | 2/107
Other Adverse Events (participants affected / at risk) | 97/141 | 97/141 | 63/108 | 57/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Type 2 Diabetes Group: Placebo + Metformin (N=141) | Type 2 Diabetes Group: Colesevelam + Metformin (N=145) | Pre-diabetic Group: Placebo (N=108) | Pre-diabetic Group: Colesevelam (N=107)
Chest pain (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Lung squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Polycystic Ovaries (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Type 2 Diabetes Group: Placebo + Metformin (N=141) | Type 2 Diabetes Group: Colesevelam + Metformin (N=141) | Pre-diabetic Group: Placebo (N=108) | Pre-diabetic Group: Colesevelam (N=107)
Abdominal distension (Gastrointestinal disorders) | 5 | 4 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 8 | 6 | 3 | 3
Abdominal pain uppper (Gastrointestinal disorders) | 3 | 5 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 6 | 5 | 10
Dyspepsia (Gastrointestinal disorders) | 5 | 5 | 0 | 3
Flatulence (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 7 | 2 | 4
Nausea (Gastrointestinal disorders) | 11 | 18 | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 6 | 0 | 3
Asthenia (General disorders) | 4 | 5 | 0 | 0
Pyrexia (General disorders) | 7 | 2 | 1 | 3
Gastroenteritis (Infections and infestations) | 3 | 2 | 0 | 0
Influenza (Infections and infestations) | 9 | 12 | 7 | 9
Nasopharyngitis (Infections and infestations) | 2 | 5 | 5 | 1
Sinusitis (Infections and infestations) | 3 | 3 | 1 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 3 | 3 | 1
Urinary tract infection (Infections and infestations) | 7 | 3 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0
Dyslipidemia (Metabolism and nutrition disorders) | 4 | 5 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 0 | 10 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 2 | 4
Dizziness (Nervous system disorders) | 5 | 9 | 0 | 5
Headache (Nervous system disorders) | 14 | 12 | 10 | 7
Somnolence (Nervous system disorders) | 3 | 2 | 0 | 0
Anxiety (Nervous system disorders) | 3 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Hypertension (Vascular disorders) | 8 | 2 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The following language is employed: "If identified by DSI, any of DSI's confidential information as defined herein shall be deleted...Nothing in this publication section shall be taken as giving DSI and right of editorial control over any publication prepared by the Study Site."